CLINICAL TRIAL: NCT06604923
Title: Advanced Molecular Imaging of Cholestatic Disorders in Humans: Pathophysiological Characterization and Treatment Effects
Brief Title: PET/CT Scans Using the Tracer 11C-Csar, a Bile Acid Analog, to Depict and Visualize Changes in the Hepatobiliary System in Patients With Primary Biliary Cholangitis Before and After Treatment.
Status: Active, not recruiting | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: Csar_PBC; 1-10-72-64-24 (Other: The Central Denmark Region Committees on Health Research Ethic)
Record Dates: First submitted 2024-09-16; First posted 2024-09-20 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Primary Biliary Cholangitis (PBC); Cirrhosis; Cholestasis; Ursodeoxycholic Acid; Bezafibrate
MeSH Terms: conditions — Liver Cirrhosis, Biliary; Fibrosis; Cholestasis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood samples in a biobank
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Purpose The primary purpose is to use an imaging diagnostic method to examine how the medication for primary biliary cholangitis (PBC) works. This will be studied using a radioactive tracer that behaves like human bile and can be observed with a PET/CT scanner. The aim is to gain insight into the disease mechanisms and how the medication affects them.

The standard treatment for PBC is ursodeoxycholic acid, also known as Ursochol, which stimulates bile flow. If treatment with Ursochol is insufficient, bezafibrate can be added. The effectiveness of treatment is currently monitored through blood tests, which do not necessarily reflect the severity of the liver disease. However, this can be assessed using advanced PET/CT scans with a radioactive tracer, 11C-CSAR, which quickly clears from the body.

The purpose of this study is to use the method to show how 11C-CSAR moves through the liver and bile ducts in PBC patients before and after treatment with either Ursochol or a combination of Ursochol and bezafibrate.

We aim to:

* Observe how the disease affects the liver&amp;amp;#39;s handling of bile salts and how this changes with medication.
* Determine the excretion kinetics of 11C-CSAR, including specific rate constants.
* Assess changes in liver blood flow before and after treatment.
* Compare routine blood tests with 11C-CSAR PET/CT findings to evaluate how well blood tests reflect actual liver involvement.

Study Plan The scientific study involves two examination days. Both days follow the same procedure. Participants must arrive fasting on the examination day. An intravenous catheter will be placed in each arm, a catheter in a wrist vessel, and a liver vein catheter. The liver vein catheter will be inserted by a trained liver doctor through a small sheath in a neck vein, guided by ultrasound, and the final placement will be confirmed with fluoroscopy. The tracer 11C-CSAR and the dye indocyanine green (ICG) will be administered through the intravenous lines. ICG will be given as a constant infusion 90 minutes before the scan to distribute in the tissue. The tracer will be injected just before the scan. Blood samples will be taken from the liver catheter and wrist catheter during the scan, which lasts approximately 45 minutes. After the scan, the catheters will be removed, and the participant can leave shortly afterward. About 250-300 ml of blood will be drawn during the scan, which will have no significant impact on participants. The entire process is expected to take about four hours.

Study Participants Our goal is to include 20 newly diagnosed PBC patients and 10 patients who do not respond to standard treatment and are about to begin bezafibrate. Some participants may complete both parts of the study. If newly diagnosed patients do not respond sufficiently to Ursochol and need to start bezafibrate while the study is ongoing, they may participate both before and after starting Ursochol and bezafibrate.

DETAILED DESCRIPTION:
Cholestasis Cholestasis is defined as decreased bile flow from the liver to the duodenum, either due to hepatocellular functional defects or obstruction of the biliary tree (1). Bile acids are essential for absorbing lipophilic compounds from the intestine (1).

The buildup of bile acids in the liver damages tissue in different ways. The bile acids disturb the movement of structural proteins within cells, change how cells maintain their polarity through internal vesicle transport, and cause irregularities in the activity of membrane transporters responsible for releasing bile (2).

Patients with cholestasis typically experience jaundice and pruritus due to bile acids accumulating in the skin. Assessing a patient with cholestasis includes a comprehensive medical history, diagnostic imaging, and laboratory analysis of blood samples. Elevated blood levels of alkaline phosphatases (ALP), gamma-glutamyl transferase, and sometimes bilirubin are observed (3).

Ultrasonography helps differentiate between intrahepatic and extrahepatic causes, with extrahepatic causes like tumours or gallstones often detectable via ultrasound, while intrahepatic causes require further investigation(1).

This study explores primary biliary cholangitis, a condition characterized by intrahepatic cholestasis.

Primary biliary cholangitis Primary biliary cholangitis (PBC; previously primary biliary cirrhosis) is an autoimmune liver disease characterized by the destruction of the intrahepatic bile ducts. The disease is more prevalent in women than men, at a ratio of 9:1 and has a chronic, progressive course potentially leading to fibrosis and cirrhosis (4). The dominant symptoms are fatigue and pruritus, negatively affecting the patient's quality of life (5). Globally, an estimated 1/1000 women above the age of 40 years live with PBC (3).

PBC may be suspected when patients have an unexplained elevation of plasma ALP without hepatobiliary obstruction. The PBC diagnosis may be established based on two of the following three criteria:

* Elevated plasma ALP,
* Detection of antimitochondrial antibodies (AMA; present in 95% of patients) or other PBC- specific autoantibodies (SP100 or GP210) in case of negative AMA,
* Non-suppurative destructive cholangitis and destruction of the interlobular bile ducts seen in liver histology (5).

The first-line treatment in patients with PBC is the bile acid analogue, ursodeoxycholic acid (UDCA)(3). UDCA stimulates bile acid metabolism by increasing hepatocyte and cholangiocyte excretion of bile acids, organic anions and biliary HCO3-(6). Treatment response is monitored by measuring ALP levels. A treatment response is defined as ALP &lt;160 U/I after one year of treatment according to the Paris II Criteria (5). Up to 40% do not respond to first-line therapy (5) and in these patients, second-line treatment with bezafibrate may be considered. Bezafibrate is a peroxisome proliferator-activated receptor (PPAR) agonist influencing bile acid synthesis. Research indicates that when combined with UDCA, bezafibrate can reduce ALP, improve symptoms, and possibly prolong the time to transplantation (5,7). However, treatment with bezafibrate is not considered standard practice and is used only in specialized centres in Denmark (8). The only treatment option for patients with advanced PBC or intolerable and treatment-resistant pruritus is liver transplantation (3).

Studying the hepatobiliary handling of bile acids has been challenging, primarily due to the liver&#39;s concealed position between the portal venous and systemic blood systems and because of the inherent difficulty in retrieving sampling materials from bile. The present project aims to quantify the functional effects of PBC treatment by non-invasive imaging of hepatobiliary excretion of bile acids using functional positron emission tomography/computer tomography (PET/CT).

Molecular imaging of cholestasis The Department of Hepatology &amp; Gastroenterology and the Department of Nuclear Medicine &amp; PET Centre, both Aarhus University Hospital, have developed a PET/CT method to study the enterohepatic circulation of bile acids. The technique utilizes the carbon-11 labelled conjugated bile acid tracer cholylsarcosine (11C-CSAR) (9-12).

11C-CSAR is a synthetic conjugate of N-methyl glycine (sarcosine) and cholic acid, which was chosen due to its similarity to taurocholic acid, one of the essential bile salts in humans. Also, this bile acid is not metabolized in the body or by bacteria in the intestines.

We have validated the 11C-CSAR PET/CT method in patients with various cholestatic disorders and healthy controls (9,11,13). We plan to enhance our dataset by utilizing newer, more advanced scanners and extending the method to include patients with primary biliary cholangitis (PBC). Currently, this method is exclusively available at Aarhus University Hospital.

Traditional monitoring of primary biliary cholangitis relies on regular blood tests for the biomarker ALP, which may not provide a comprehensive understanding of disease progression. Additionally, there&#39;s uncertainty about why certain patients don&#39;t respond to treatment, and existing clinical tools fail to predict treatment outcomes reliably. Common imaging modalities lack the specificity needed for detailed evaluation. Expanding our methodological approach and access to more advanced imaging technology will potentially address these limitations and improve patient care.

This study aims to quantify the changes in the in vivo hepatobiliary secretion kinetics before and after standard treatment with 1) UDCA in treatment-naïve patients with PBC and 2) bezafibrate as an add- on treatment in patients with PBC who are non-responders to UDCA. The study will apply functional hepatobiliary PET/CT imaging using the conjugated bile acid tracer 11C-CSAR. The study will generate new knowledge about the pathophysiological background of PBC and demonstrate how and where the medicine works. To quantify these changes in the in vivo hepatobiliary secretion kinetics, we scan the same patients twice.

Study design Patients need to come twice to quantify these changes. The study is an investigator-initiated, exploratory, observational study of patients with PBC, conducted before and after standard treatment with UDCA alone or combined with bezafibrate. It consists of two study arms: 1) treatment-naïve patients newly diagnosed with PBC who initiate standard treatment with UDCA, and 2) patients with PBC who are non-responders to UDCA and initiate second-line treatment with bezafibrate. Some patients are thus investigated twice after the baseline scan and diagnosis since only non-responders to UDCA patients are offered second-line treatment with bezafibrate according to guidelines.

The study starts at 8.00 AM after an overnight fast. The participants will have catheters placed in the hepatic vein, two peripheral veins and a radial artery for blood sampling. Indocyanine green (ICG) will be administered intravenously in a vein to measure hepatic flow (Fick&#39;s principle).

The radiotracer 11C-CSAR is administered intravenously at the beginning of a 45-minute PET/CT scan. Blood samples will be drawn from the arterial and hepatic vein catheter during the scan to measure hepatic blood flow and 11C-CSAR concentrations during the scan. ALP and bile salts will also be measured from the blood.

Methods 11C-CSAR PET/CT 11C-CSAR is injected intravenously in micro-doses at the beginning of a dynamic PET/CT scan of the biliary system. The radiotracer is taken up by the hepatocytes and secreted into the intestine through the bile duct (9-13). By continuous external recording, the PET camera provides real-time measurements of the time course of tissue concentrations of 11C-CSAR in liver tissue, bile ducts, etc.

The 11C-CSAR PET/CT scans are performed after an overnight (8-hour) fast. The participants are placed in a supine position in the (Siemens Quadra) with the liver within the 21cm field of view. A low-dose CT scan is used to visualize the anatomy. 25-50 MBq 11C-Csar dissolved in 10 ml of saline water is administered intravenously as a 25-second bolus at the beginning of a 45-minute PET/CT scan. During the scan, blood samples from the hepatic vein catheter are drawn to measure concentrations of 11C- CSAR.

Venflons are placed percutaneously in both cubital veins by a trained technician for intravenous administrations of 11C-CSAR and ICG. For blood sampling, an arterial catheter (Artflon) will be percutaneously placed in the radial artery by a trained anesthesiologist, and a catheter will be inserted into the hepatic vein via the right jugular vein by a trained hepatologist. The insertion is guided by ultrasound sonography using local anaesthesia and an aseptic technique. The catheter placement will be verified via fluoroscopy.

Blood samples Patients undergo blood sampling in their standard treatment program to assess disease progression and general health status. This includes tests for liver enzymes (ALT, AST), bilirubin, ALP, albumin, PT/INR, ammonium, amylase, lipid profile, glucose, HbA1c, TSH, haemoglobin, platelets, CRP, soluble (s)CD163, and white blood cells with differential count. Potassium, sodium, creatinine, eGFR, calcium metabolism, thyroid function, and total cholesterol are often also measured. The blood is discarded immediately after analysis.

11C-CSar blood concentrations, ICG blood concentrations and ALP are determined immediately, and the blood is disposed of afterwards. Blood for plasma bile salt concentrations is stored in a freezer and analyzed collectively after the last participant has been included. Any remaining plasma is destroyed immediately after analysis.

If the patient accepts this, 30 ml of blood is stored in the research biobank for 15 years (see below).

Data analysis The data comprise 11C-CSAR concentrations in liver and bile ducts (PET data) and arterial and hepatic venous blood concentrations of 11C-CSAR and hepatic blood flow calculated from ICG (Ficks principle). These data are used to calculate kinetic rate constants for uptake from sinusoidal blood into hepatocytes (ml blood/min/ml liver tissue), back-flux to sinusoids (/min), transport from hepatocytes into biliary canaliculi (/min), and bile flow (ml bile/min). Mean transit time in hepatocytes (min) and relative tissue concentrations are also calculated (9-13).

Data Management Source data for each participant is registered in the participant's PET journal or Case Report Form (CRF). The CRF is established as a project in REDCap and contains information on contact information and demography (sex, weight, height).

The PET journal contains all data, including tracer production, quality control, administered dose, and scan data (including possible deviations and complications). The localization of source data is kept in the trial master file (TMF). The signed consent forms are kept in digital form in REDCap, and a physical form is kept in a locker with the TMF. Data is held in the eCRF (REDCap) and the PET journal.

All research participants will perform data analysis and management.

Sample size and statistics We plan to include 20 patients with PBC before and after UDCA and ten patients before and after bezafibrate. Our experience from similar studies shows that this number of patients is appropriate for a paired PET/CT examination like this one(9,11,13). Previous studies have demonstrated significant differences between healthy individuals and patients. When patients begin treatment with ursodeoxycholic acid (UDCA), some expect to achieve normal alkaline phosphatase levels, assuming no cholestasis. In previous experiments, we have observed changes in the rate at which the tracer moves from the hepatocyte to the intrahepatic bile duct, from 0.12 minutes in patients to 0.41 minutes in healthy participants.

n1= >miredif2 (z1-2alfa+z1-beta) x SD2 MIREDIF (Minimum Detectable Difference): The observed difference between the rate at which a tracer moves from the hepatocyte to the intrahepatic bile duct before and after treatment is 0.29 minutes. Standard Deviation (SD) The variability in our data ranges from 0.01 to 0.51 minutes.

Significance Level (alfa): Set at 0.05, representing the threshold for statistical significance.

Power (1-beta)Set at 0.8, indicating the probability of detecting an actual effect if it exists.

n! > (1,96 + 0,84)x 0,51 =n! = 8,6 Calculations confirm that 9 participants in each group would be sufficient to obtain reliable results in our study. Considering potential dropout rates and to ensure robustness in our analysis, we will recruit a slightly larger number of participants than the calculated minimum.

Statistical analyses are performed in STATA 16/18 and GraphPad Prism 9.0 in pseudonymized form. Data are deleted or anonymized after ten years.

Data are analyzed per protocol, and participants who withdraw from study treatment or have missing data regarding the primary endpoints will be excluded from the analysis. The results will state if any deviations from the statistical analysis plan occur. Should a participant withdraw from the study before completion, a new participant will be recruited to ensure we have a complete dataset of participants.

Paired endpoint changes will be statistically tested using the paired t-test or the Signed rank test in case of non-normally distributed or skewed data. Correlations between endpoints will be tested using the Pearson or Spearman correlation coefficients in case of non-normally distributed or skewed data.

Risk, side effects and precautions

Monitoring during and after 11C-CSAR PET/CT During 11C-CSAR PET/CT, participants are under constant medical supervision. The Department of Nuclear Medicine & PET Centre has all the necessary equipment and medication in case of acute tracer- related reactions. We do not anticipate any allergic reactions as the tracer 11C-CSAR acts like taurocholic acid, an endogenous human bile salt, and it is administered in tracer dose. The ICG poses a minimal risk of allergic reactions. The personnel monitoring the participants are trained in treating a critical allergic response. Any reactions will be monitored closely and reacted upon.

All catheters are removed after the 11C-CSAR PET/CT scan, and the participants can leave 30 minutes later. All participants are encouraged to contact us if they feel discomfort or have concerns regarding the trial and the scans after participating.

Radiation risk The 11C-CSar dose used for each PET scan is 0,5 MBq/kg with a minimum of 25 MBq and a maximum of 50 MBq. The effective radiation dose of 11C-Csar is 0,0062 mSv/MBq(15). An average person weighing 75 kg is thus exposed to 0,23 mSv from one 11C-Csar PET/CT scan. The radiation dose from the low-dose CT scan is 2,3 mSv. The total radiation exposure from 2 11C-CSar PET/CT scans is accordingly (2*0,23 + 2*2,3) = 5 mSv.

As per appendix II "Retningslinjer om anvendelse af ioniserende stråling i sundhedsvidenskabelige forsøg", this corresponds to the risk category IIb. Compared to the annual background radiation, which is 3 mSv, the given value of 5 mSv represents a relatively small contribution.

The general 25% lifetime cancer risk is increased to 25.025% for a patient participating in the study.

Non-responders to first-line treatment will have the opportunity to participate after starting second- line treatment with bezafibrate. These patients may undergo up to three 11C-Csar scans during the study period, although the number of these patients is expected to be low. If they undergo three 11C- Csar scans, their radiation exposure will be 7,59 mSv and still fall within category IIb.

This corresponds to approximately three years of background radiation and increases their lifetime cancer risk to 25.38%.

Information from medical records 11C-CSAR is a synthetic conjugate of N-methyl glycine (sarcosine) and cholic acid, which we chose due to its similarity to taurocholic acid, one of humans' essential bile salts. No adverse events have previously been observed.

ICG is a routine test for measuring hepatic flow, and adverse events are infrequent.

Insertion of the catheters may cause a small amount of pain, subcutaneous bleeding and pose a minimal risk of superficial infection. These catheters are used daily in the hospital without any side effects.

Inserting a hepatic vein catheter carries a risk of bleeding, thrombosis and infection. In our clinic, the occurrence of these side effects is less than 1/1000. The procedure is performed routinely about 120 times a year for clinical investigations, and we have yet not experienced any complications.

During the 11C-CSAR PET/CT scan, blood samples from the participants are collected from the artflon in the radial artery and the hepatic vein catheter. In total, 250 - 300 ml of blood is drawn from the participants. This blood loss is of no risk for the participants.

The investigator will review information from the electronic medical records (Midt-EPJ) regarding patients listed on the outpatient lists and admission in the bed wards (fulfilment of in- and exclusion criteria) before obtaining informed consent, and the information will be passed on to the project afterwards. This information has been disclosed to the investigator from the medical records. Before obtaining informed consent, information from about 75 patients will be passed on to the investigator. This information is based on records from the past five years. Information from the participating patient's medical charts will be collected for the project from all 30 patients after obtaining written, informed consent. The informed consent gives the investigator and the investigator representatives direct access to information about the study participants' health status from their electronic medical patient records. The data includes gender, age, medical history, current medication, biopsy results, pathology reports and biochemical test results.

Respect for the physical and mental integrity and the privacy of the study participants The consent provides the investigators, their representatives, and any regulatory authority direct access to obtain information from the patient's medical records, including electronic records, to review the study participant's health status necessary for the implementation of the research project and for monitoring purposes, including self-inspection, quality control, and monitoring, which they are obligated to perform.

All data will be treated confidentially and according to the applicable Danish legislation.

When participants have signed a consent, information from their health records will be collected, according to §43, 1 in the Danish Health Law. This information includes sex, age, height, weight, blood tests, other diseases, imaging such as ultrasound sonograph, liver biopsy, and other medication. Access to this information will be used to evaluate and monitor the study and determine participants' general health and liver function. The information will be used in the scientific publication of the study results and will be fully anonymized so that no personally identifiable data will be published. Information regarding the participants will be protected according to the General Data Protection Regulation (GDPR), the Data Protection Act, and the Danish Health Law §43 will be complied with.

Biobank for further research The participants are informed that a biobank is established with the possibility of conducting additional analyses related to primary biliary cholangitis and that they can participate in the project without donating blood to the biobank. If they accept to donate blood, approximately 30 ml of blood is stored in the biobank. The material will be stored for up to 15 years, and if we wish to utilize the material, approval will be sought from the Regional Ethics Committees for Region Midt. Patients may request the destruction of their material in the biobank at any time. Blood stored in the biobank will be protected according to the General Data Protection Regulation (GDPR) and the Data Protection Act.

Financial statement The involved scientists initiated the study, and none of the involved partners have any economic interests in the study. The project is financed by Novo Nordisk Fonden (1 mil. DKK of 8.506500,00 DKK). The grant is provided for a more extensive research program on liver disease and imaging modalities (given to Michael Sørensen). The expenses include the salary for PhD student Maja Kanstrup Jørgensen and all expenses regarding the study, including but not limited to scans, blood samples, and compensation to the participants.

Reimbursement Recruitment of participants The patients will not receive reimbursement, but we will cover documented travel expenses, overnight stays at the patient's hotel, and documented lost wages.

When a patient who meets the inclusion criteria is admitted to the departments or comes in for an outpatient visit, the doctor who sees the patient will inform about the opportunity to take part in the study and ask for permission for an investigator to see or call the patient with initial information about the study and to arrange for a physical meeting and conversation about the study. If the patient accepts this, ID and contact information are given to Maja or an investigator representative, who then contact the patient for oral information about the project. Maja or the investigator representative will also make sure (from the electronic patient file) that the patient meets the inclusion criteria and none of the exclusion criteria. If the patient continues to show interest in the study, the written project information and the brochure "Forsøgspersons rettigheder i et sundhedsvidenskabeligt forskningsprojekt" will be handed out or sent via Eboks.

When the patient has read the material, the primary investigator, Maja, or an investigator representative will have an in-depth discussion with the participant about the nature of the study and the rights of the study subject. The participant will be informed about the right to bring an assessor, and how the consent can be withdrawn at any time without reason. The conversation will occur in quiet surroundings with enough time to discuss the study thoroughly. The investigator will ensure the participant understands the study and inform them of their right to consider participation for at least 24 hours before consenting.

Written and verbally informed consent will be obtained before participation in the study can begin. Information about the possibilities of complaint and possible compensation regarding unforeseen side effects is given.

Publication of the results All positive, negative, or inconclusive results will be published. Results will be presented at Danish and international meetings and published in international peer-reviewed scientific journals with author lists according to the ICMJE recommendations.

Ethical aspects of the study The tests are carried out under the principles of the Helsinki Declaration II with appendix after approval by The Committee on Health Research Ethics for Region Midt. Inclusion of participants follows the ethical guidelines set out by The Ethics Committee on request upon participation, obtainment of informed consent, information on trial subjects' rights, etc.

11C-CSAR PET/CT has been used several times in patients and healthy individuals in the department without any adverse events. As mentioned, the tracer 11C-CSAR has no therapeutical effect and is not metabolized.

Participation in the study does not directly benefit the individual patient, but the results will hopefully increase our pathophysiological knowledge of patients with primary biliary cholangitis. Participation will have no impact on standard treatment.

In our opinion, the risks and possible side effects are outweighed by the expected benefits.

When signing the informed consent letter, participants will decide if they want information on unexpected findings in the scans. Should incidental results occur during the scans, the participants will be informed and offered regular clinical examinations.

Criteria for interruption of the study for each patient Criteria for interruption of the study - Unexpected severe adverse events related to the study in more than one participant.

Insurance

"Patienterstatningen" will cover subjects if necessary.

* The participant withdraws the consent.
* The responsible physician considers the participant's health endangered by continuing the trial.

Timeline Inclusion will start shortly after approval from The Committee on Health Research Ethics for Region Midt. PET/CT scans will be planned weekly when the patients are in the departments. The project is terminated after the last scan is completed or no later than five years after the approval of the study. Data management will be performed concurrently and finished within the duration of the project

ELIGIBILITY:
Inclusion Criteria:

* - A clinical diagnosis of PBC as defined by guidelines (3).
* Age ≥ 18.
* For fertile female participants: A negative urinary pregnancy test performed on the day of the scan.
* Treatment-naïve patients:

  * DiagnosisofPBCwithin<1year
  * NopriortreatmentforPBC(UDCA,bezafibrate)
* Non-responders to UDCA:

  * Insufficient treatment response to UDCA defined by guidelines (ALP>160U/I)

Exclusion Criteria:

* - Pregnancy
* Claustrophobia or the inability to remain still during a 45-minute scan.
* Coagulation deficiency that does not allow hepatic vein catheter (relative).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with primary biliary cholangitis from The Central Region in Denmark,
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-09-04 (Actual); Primary Completion 2029-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
The aim of this study is to apply the 11C-CSAR PET/CT method to quantify hepatobiliary secretion kinetics of 11C-Csar in patients with primary biliary cholangitis before and after treatment | through study completion, an average of 2 years
  - Changes in the hepatobiliary excretion kinetics of 11C-CSar after treatment with 1) UDCA or 2) UDCA and bezafibrate

SECONDARY OUTCOMES:
Aim The aim of this study is to apply the 11C-CSAR PET/CT method to quantify hepatobiliary secretion kinetics of 11C-Csar in patients with primary biliary cholangitis before and after treatment | Through study completion, an average of 2 years
  - Changes in hepatic blood flow (L/min) after 1-4 months of treatment with 1) UDCA or 2) Bezafibrate.
The aim of this study is to apply the 11C-CSAR PET/CT method to quantify hepatobiliary secretion kinetics of 11C-Csar in patients with primary biliary cholangitis before and after treatment | Through study completion, an average of 2 years
  - Changes in blood markers of cholestatic liver injury (ALP and other clinically used blood tests) after treatment with 1) UDCA or 2) UDCA and bezafibrate.)

CONTACTS AND LOCATIONS:
Locations (1):
- The Department of Hepatology and Gastroeneterology Aarhus University Hospital., Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Undecided